CLINICAL TRIAL: NCT07098299
Title: A Phase I Dose-escalation and Metabolomics Study of Metformin Combined With Chemotherapy and/or Immunotherapy in Solid Malignancies
Brief Title: Metformin Combined With Chemotherapy and/or Immunotherapy in Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Wasif Saif, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-050
Record Dates: First submitted 2025-07-10; First posted 2025-08-01 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Metformin will be administered in combination with any standard chemotherapy/immunotherapy. Metformin 1000mg-3000mg day in dose escalation
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be given for 14 days alone as a run in and then added to any standard of care chemotherapy or immunotherapy for solid tumors.

SUMMARY:
The goal of this clinical trial is to evaluate the safety of Metformin alone and in combination with chemotherapy or immunotherapy in patients with solid tumor cancers. The main questions it aims to answer are:

* what are the toxicities of metformin at multiple dose levels
* what is the maximum tolerated dose of Metformin in combination with chemotherapy or immunotherapy

Participants enrolled will be treated with standard of care chemotherapy and/or immunotherapy in accordance to their disease/stage. In addition, participants will take Metformin alone for 14 days in between the first cycle of chemotherapy and the second cycle of chemotherapy to determine tolerability to the Metformin. Participants will then take Metformin daily in combination with the standard of care chemotherapy and/or Immunotherapy from cycle 2 onwards.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed advanced solid tumor and are considered a suitable candidate for chemotherapy and/or immunotherapy or both
* Are a male or female participant aged ≥ 18 years
* Have provided a signed, written informed consent form
* Have measurable disease per RECIST v1.1
* Have adequate hematologic, renal, liver, and coagulation function as defined by the following:

  1. Hemoglobin ≥ 8 g/dL if determined suitable by the investigator for the selected chemotherapy and/or immunotherapy regimen for the particular patient
  2. Absolute neutrophil count (ANC) > 1500/mm3
  3. Platelets > 75,000/mm3 if determined suitable by the investigator for the selected chemotherapy and /or immunotherapy regimen for the particular patient
  4. Estimated Glomerular Filtration Rate (eGFR) > 45 mL/min/1.73 m2 (as described by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] 2021 equation)
  5. Total bilirubin ≤ 1.5 x upper limit of normal (ULN). Participants with known Gilbert's syndrome who have total bilirubin level ≤ 3 x ULN may be enrolled if deemed suitable for a particular patient by the investigator for the selected chemotherapy and/or immunotherapy regimen.
  6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN. For participants with hepatic metastases, AST and ALT ≤ 5 x ULN.
  7. Alkaline phosphatase (ALP) < 2.5 x ULN. For participants with hepatic and/or bone metastases ≤ 5 x ULN
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2, and suitable for chemotherapy/IO recommended by the investigator.
* Participants who have experienced expected toxicity from Cycle 1 of anticancer therapy which is unlikely to recover to grade 1 or better prior to Cycle 2 (e.g., anemia, alopecia, vitiligo, endocrine dysfunction associated with IO) and may otherwise not impact the eligibility will be allowed.
* Women of child-bearing potential must agree to avoid becoming pregnant and male participants should avoid impregnating a female partner or donating sperm starting at initiation of treatment up until at least 90 days after the last dose of study drug.
* Have an estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Patients who have or are any of the following exclusion criteria are not eligible for participation in the study.
* Patients with uncontrolled diabetes
* Patients who have received metformin must be at least five half-lives beyond such treatment (four weeks) and must not be taking metformin at the time of enrollment.
* Patients with a known hypersensitivity to metformin, its excipients, its analogs, or any of its components
* Patients on other antidiabetic medicines are eligible as long as adding metformin will not be contraindicated
* Patients with an inability to tolerate oral medications
* Women who are pregnant or lactating
* Patients with clinically significant intercurrent disease including, but not limited to:

  1. New York Heart Association Class III or IV heart failure
  2. Myocardial infarction, unstable angina, or stroke ≤ 3 months prior to Cycle 1 Day 1
  3. Uncontrolled arrhythmia
  4. Clinically significant active infection requiring IV antibiotic, antiviral, or antifungal medications
* Patients with other current medical or other conditions that, in the opinion of the investigator, may confound study interpretation or prevent completion of study procedures and follow-up examinations
* Patients with an unwillingness or inability to comply with the study procedures required in this protocol
* Patients using an investigational agent within four weeks of study entry
* Patients with uncontrolled metabolic disorders or primary or secondary effects of cancer that induce a high medical risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-07-07 (Estimated); Study Completion 2028-07-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs)-Metformin only stage | From the start of Metformin run in to the end of Metformin run in. Up to 14 days
  Adverse events (AEs) and serious adverse events (SAEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0).
Incidence of Dose Limiting Toxicities (DLTs)-Chemotherapy or Immunotherapy (IO) plus Metformin Stage | From start of Chemotherapy or IO plus Metformin until 30 days after the end of treatment
  Adverse events (AEs) and serious adverse events (SAEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0).
Determine the maximum tolerated dose (MTD) of metformin in combination with chemotherapy/IO | Up to 4 months after treatment initiation
  The MTD will be defined as the dose level below the dose level at which two or more patients in the same cohort experience a DLT. If none or only one patient experiences a DLT at level 5, then dose level 5 will be defined as the MTD.

SECONDARY OUTCOMES:
Assessment of overall response rate (ORR) | Up to 4 months after treatment initiation
  Tumor response will be determined according to RECIST v1.1. Treatment responses will be summarized by count and percentage, and their rates will be computed along with their associated two-sided 95% confidence intervals (CIs).
Assessment of Duration of Response (DOR) | Up to 4 months after treatment initiation
  Tumor response will be determined according to RECIST v1.1. The DOR is measured from the time measurement criteria are met for complete response (CR) or a partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started). Treatment responses will be summarized by count and percentage, and their rates will be computed along with their associated two-sided 95% confidence intervals (CIs). The distributions of time-to-event data, such as DOR and PFS will be graphically summarized using Kaplan-Meier (KM) curves, and their median and 95% CIs will be estimated using KM estimates.
Assessment of Progression free survival (PFS) | Up to 4 months after treatment initiation
  Tumor response will be determined according to RECIST v1.1. Progression-free survival (PFS) is defined as the time duration from treatment start to progression time or death, whichever occurs first. Treatment responses will be summarized by count and percentage, and their rates will be computed along with their associated two-sided 95% confidence intervals (CIs). The distributions of time-to-event data, such as DOR and PFS will be graphically summarized using Kaplan-Meier (KM) curves, and their median and 95% CIs will be estimated using KM estimates.

OTHER OUTCOMES:
Evaluate extracellular nicotinamide phosphoribosyltransferase (eNAMPT) as a surrogate marker for nicotinamide adenine dinucleotide (NAD) signaling inhibition | Up to 4 months after treatment initiation
  Serum NAD+ and eNAMPT will be measured at baseline and every 8 weeks after the start of metformin. Enzyme linked immunosorbent assays (ELISAs) will be used to determine levels. Summary statistics (numerical and/or graphical) for changes of NAD+ and eNAMPT levels between baseline and after treatment will be evaluated, along with their summaries at the baseline and at after treatment. Correlations between NAD+ and eNAMPT to the ORR, DOR, and PFS will be calculated from patients who have a partial (at least a 30%) complete response to treatment.
Assess metabolic parameters | Up to 4 months after treatment initiation
  Glycated hemoglobin, glucose, insulin, Insulin like growth factor-1, and C-peptide levels will be measured at baseline and every 8 weeks after the start of metformin. Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated at the same timepoints. Summary statistics (numerical and/or graphical) of the metabolic parameters will be evaluated at baseline and every 8 weeks. Comparing the pretreatment biomarker levels with the post treatment levels to determine the effect of the drug using Wilcoxon signed rank test. The differences between the responding and non-responding groups using Wilcoxon-Mann-Whitney test for statistical significance will also be compared. The correlation of the metabolic parameters with tumor markers and efficacy (ORR, DOR, and PFS) will be assessed using Pearson correlation and scatter plots.
Perform metabolomics analysis | Up to 4 months after treatment initiation
  Blood will be drawn at baseline and every 8 weeks after the start of treatment. Using Liquid Chromatography Tandem Mass Spectrometry (LC-MS/MS) and MetaboAnalyst, a panel of over 200 polar metabolites will be investigated and their correlation with metformin responsiveness and PFS will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wasif Saif, M.D., Principal Investigator — Wayne State University
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States